CLINICAL TRIAL: NCT01097603
Title: L&T Noninvasive Blood Pressure Module Performance Validation
Brief Title: Larsen & Toubro (L&T) Noninvasive Blood Pressure Module Performance Validation
Status: Completed | Type: Observational
Sponsor: Larsen & Toubro Limited (Industry)
Responsible Party: L&T MEDICAL EQUIPMENTS & SYSTEMS, MYSORE,INDIA, LARSEN & TOUBRO LIMITED
Other Study IDs: LTMED01-0310
Record Dates: First submitted 2010-03-31; First posted 2010-04-01 (Estimated); Last update posted 2010-04-01 (Estimated); Status verified 2010-03

CONDITIONS: Blood Pressure
Keywords: Non-Invasive Blood Pressure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
To validate accuracy of the readings of noninvasive blood pressure (NIBP) module with sphygmomanometer as per the requirements of AAMI SP10:2002. This study is for adult and pediatric population.

ELIGIBILITY:
Subjects: Healthy volunteers

Inclusion Criteria:

* Healthy subjects
* Age between 1 - 60 yrs
* Both genders
* Consenting for the study

Exclusion Criteria:

* Subjects suffering from cardiorespiratory, neurological or endocrinal disorders
* Subjects with alcohol abuse/dependance
* Female subjects who are pregnant or lactating
* Subjects with pace maker implantations

Subjects: Diseased subjects

Inclusion Criteria:

* Patients of hypertensive, ICU and in patients of different diseases
* Age between 1 - 80 yrs
* Both genders
* Consenting for the study

Exclusion Criteria:

* Healthy volunteers

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Total 92 numbers of subjects or patients were studied during this study.
Sampling Method: Non-Probability Sample